CLINICAL TRIAL: NCT04645368
Title: Multicenter, Open-label Prospective Cohort Study of the Efficacy and Safety of the Inclusion of Longidaze in the Prevention and Treatment of Post-inflammatory Pulmonary Fibrosis and Interstitial Lung Diseases Caused by COVID-19.
Brief Title: Study of Longidaze in the Prevention & Treatment of Pulmonary Fibrosis, Interstitial Lung Diseases Caused by COVID-19
Status: Completed | Type: Observational
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Other Study IDs: DISSOLVE
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Fibroses, Pulmonary
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Longidaze: 80 subjects Longidaze® (bovhyaluronidase azoxymer), lyophilisate for solution for injection
  Interventions: Drug: bovhyaluronidase azoxymer
- Dynamic control: 80 subjects Patients not receiving active therapy

INTERVENTIONS:
Drug: bovhyaluronidase azoxymer — 3000 IU intramuscularly once every 5 days with a course of 15 injections
  Other Names: Longidaze
  Groups: Longidaze

SUMMARY:
A study is being conducted to evaluate the efficacy and safety of Longidaze for the prevention and treatment of post-inflammatory pulmonary fibrosis and interstitial lung disease following COVID-19.

DETAILED DESCRIPTION:
The aim of the study is to compare the outcomes associated with postinflammatory pulmonary fibrosis and interstitial lung disease among a cohort of adult patients after complicated pulmonary manifestations of COVID-19 in two groups: in a group of patients who were prescribed Longidaze® for treatment or prevention as part of routine clinical practice, and in the group of patients who underwent dynamic observation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with residual lung changes after complicated COVID-19
2. Residual changes were detected no later than 2 months after the discharge after disease
3. Treatment of COVID-19 was in accordance with the standard of the then current temporary guidelines for the treatment of COVID-19
4. Age of patients over 18 years old
5. Negative polymerase chain reaction (PCR) test COVID-19 at least 2 times in respiratory samples or based on serology results in blood samples
6. Patients in the framework of routine clinical practice, in accordance with the instructions for use before inclusion in the study, were prescribed intramuscular treatment with Longidaze® at a dose of 3000 IU, 1 injection every 5 days for a total course of 15 injections or dynamic observation without the use of active therapy
7. The patient did not participate in other drug clinical trials within 1 month prior to Visit 1.
8. The patient or patient's caregiver agrees to participate in the trial and sign an informed consent form
9. Patient understands and agrees to follow the planned procedures.
10. Women with fertile potential must agree to use at least one method of contraception before completing participation in the study.

Exclusion Criteria:

1. Women during pregnancy and lactation and women planning to become pregnant during the study period
2. Severe background diseases, such as severe heart failure (class IV heart function), severe liver and kidney disease, severe bronchial asthma, severe chronic obstructive pulmonary disease, bronchiectasis, bullous emphysema and previously identified interstitial lung diseases, neurological diseases, tumors.
3. Long-term bed rest, regardless of its cause
4. Increased individual sensitivity to the components of the studied drug
5. Pathological conditions that determine the impossibility of patient participation in the study (by the decision of the investigator)
6. Medical history that, according to the investigator, does not allow the patient to be included in the study
7. A burdened allergic anamnesis, which, according to the investigator, does not allow the patient to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (over 18 years old) with residual changes in the lungs against the background of the transferred COVID-19, who were prescribed Longidaze®, lyophilisate for solution for injection, 3000 IU or underwent dynamic observation without the use of active therapy
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
The severity of lung tissue lesions with fibrosis and interstitial changes on day 75 | Day 0, Day 75
  The severity of pulmonary tissue lesions with fibrosis and interstitial changes (%) according to high resolution computed tomography examination relative to the baseline value after 2.5 months in patients of the Longidaze® group compared with the dynamic observation group according to the results of a blinded central laboratory

SECONDARY OUTCOMES:
The severity of lung tissue damage by fibrosis and interstitial changes (%) on day 180 | Day 0, Day 180
  The severity of lung tissue damage by fibrosis and interstitial changes (%) according to high resolution computed tomography examination relative to the baseline value after 6 months in relation to the baseline values of the indicator in patients of the Longidaze® group in comparison with the the dynamic observation group (according to the results of a blinded central laboratory)
The severity of lung tissue lesions with fibrosis and interstitial changes (%) on day 75 and day 180 | Day 0, Day 75, Day 180
  The severity of lung tissue lesions with fibrosis and interstitial changes (%) according to high resolution computed tomography examination relative to the baseline value after 2.5 months and 6 months in patients of the Longidaze® group compared with the the dynamic observation group (according to the results of the local laboratory)
The severity of lesions of the lung tissue with fibrosis and interstitial changes and indicators: frosted glass, hydrothorax, consolidation (%) images analyzed by the Botkin.AI program (artificial intelligence) | Day 75, Day 180
  The severity of lesions of the lung tissue with fibrosis and interstitial changes and indicators: frosted glass, hydrothorax, consolidation (%) based on the high-resolution computed tomography images analyzed by the Botkin.AI program (artificial intelligence) and then verified by a specialist after 2.5 months and 6 months from the beginning of observation in relation to the baseline values of indicators in patients of the Longidaze® group in comparison with the dynamic observation group
Change in forced vital capacity (FVC) | Day 0, Day 75, Day 180
  Change in forced vital capacity FVC (%) relative to the baseline value after 2.5 months and 6 months in patients of the Longidaze® group compared with the the dynamic observation group
Change in the diffusion capacity of the lungs | Day 0, Day 75, Day 180
  Change in the diffusion capacity of the lungs (%) relative to the baseline value after 2.5 months and 6 months in patients of the Longidaze® group compared with the the dynamic observation group
Change in the degree of dyspnea on the MMRC scale | Day 0, Day 75, Day 180
  Change in the degree of dyspnea on the MMRC scale from baseline after 2.5 months and 6 months in patients of the Longidaze® group compared with the dynamic observation group.
  MMRC scale (Modified Medical Research Council scale) 0 - no - Dyspnea does not bother, except for very intense exercise
  1. - mild - Shortness of breath bothers with brisk walking or climbing a small elevation
  2. - moderate to severe - Shortness of breath results in slower walking compared to other people of the same age, or need to stop while walking at normal pace on a level surface
  3. - Severe - Shortness of breath makes you stop when walking about 100 m or after a few minutes of walking on a flat surface
  4. - very severe - Shortness of breath makes it impossible to leave the house or appears when dressing and undressing
Changes in capillary blood oxygen saturation (SpO2) | Day 0, Day 75, Day 180
  Changes in SpO2 of capillary blood relative to the initial value after 2.5 months and 6 months in patients of the Longidaze® group compared with the dynamic observation group.
Changes in the covered footage in the 6-minute walk test | Day 0, Day 75, Day 180
  Changes in the covered footage in the 6-minute walk test after 2.5 months and 6 months in patients of the Longidaze® group compared with the dynamic observation group.
Changes in capillary blood saturation (SpO2) after a 6-minute walk test | Day 0, Day 75, Day 180
  Changes in capillary blood saturation (SpO2) after a 6-minute walk test after 2.5 months and 6 months in patients of the Longidaze® group compared with the dynamic observation group.
Change in the residual volume of the lungs | Day 0, Day 75
  Change in the residual volume of the lungs after 2.5 months in patients of the Longidaze® group compared with the dynamic observation group.
Change in the total lung capacity | Day 0, Day 75
  Change in the total lung capacity after 2.5 months in patients of the Longidaze® group compared with the dynamic observation group.
Change in inspiratory capacity | Day 75
  Change in inspiratory capacity after 2.5 months in patients of the Longidaze® group compared with dynamic observation group

CONTACTS AND LOCATIONS:
Locations (15):
- Russia (15):
  - Federal State Budgetary Educational Institution of Higher Education "Astrakhan State Medical University" of the Ministry of Health of the Russian Federation, Astrakhan, Astrakhan Oblast
  - Municipal autonomous health care institution "City Clinical Polyclinic No. 8", Chelyabinsk, Chelyabinsk Oblast
  - State Budgetary Healthcare Institution "Regional Clinical Hospital No. 3", Chelyabinsk, Chelyabinsk Oblast
  - Municipal budgetary institution "Central city clinical hospital number 6 ", Yekaterinburg, Ekaterinburg Region
  - Medical center "Clinic South", Krasnodar, Krasnodarskiy Kray
  - Federal State Budgetary Scientific Institution "Federal Research Center" Krasnoyarsk Scientific Center of the Siberian Branch of the Russian Academy of Sciences " Scientific Research Institute of Medical Problems of the North, Krasnoyarsk, Krasnoyarsk Region
  - Institute of Clinical Immunology LLC, Krasnoyarsk, Krasnoyarsk Region
  - St. Petersburg State Budgetary Healthcare Institution "City Consultative and Diagnostic Center No. 1", Saint Petersburg, Leningradskaya Oblast'
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk, Novosibirsk Oblast
  - CJSC "Medical Center" Philosophy of Beauty and Health ", Perm, Perm Krai
  - State budgetary institution of health care Republican clinical hospital named after G.G. Kuvatova, Ufa, Ufa Region
  - State health care institution "Clinical Hospital No. 4", Volgograd, Volgograd Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Volgograd State Medical University" of the Ministry of Health of the Russian Federation Volgograd State Medical University of the Ministry of Health of Russia, Volgograd, Volgograd Oblast
  - FSBI "Main Military Clinical Hospital named after Academician N.N.Burdenko" of the Ministry of Defense of the Russian Federation, Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow "City Polyclinic No. 180 of the Department of Healthcare of the City of Moscow", Moscow

IPD SHARING:
Plan to Share IPD: No